CLINICAL TRIAL: NCT02818465
Title: Role of the Interaction Between AGEs and Their Receptor RAGE in the Development and the Progression of the Uremic Vasculopathy of Hemodialyzed Patients
Brief Title: Role of the Interaction Between Advanced Glycation End Products and Their Receptor RAGE in the Development and the Progression of the Uremic Vasculopathy of Hemodialyzed Patients
Acronym: RAGE-VASCU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PR14037
Record Dates: First submitted 2016-06-23; First posted 2016-06-29 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2018-04

CONDITIONS: Hemodialyzed Patients

ARMS (1):
- Patients (Experimental)
  Interventions: Other: Vascular calcifications by Xray; Other: Vascular calcifications by tomodentimetry; Biological: Blood sample withdrawn

INTERVENTIONS:
Other: Vascular calcifications by Xray
Other: Vascular calcifications by tomodentimetry
Biological: Blood sample withdrawn

SUMMARY:
Chronic kidney disease (CKD) is associated with an extensive vasculopathy and high cardiovascular mortality as well as an accumulation of uremic toxins. Among the latest, advanced glycation end-products (AGEs) interact with RAGE. Investigators aimed to analyze the role of RAGE in the calcification process of hemodialyzed patients, in a correlative and prospective study. Vascular calcifications will be assessed by Xray and tomodentimetry while accumulation of AGEs will be measured in the serum and in the skin (non invasive). Additionally factors influencing RAGE activation such as genetic polymorphism and level of soluble forms of RAGE will be measured and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Renal impairment
* Hemodialysis for more than 3 months
* Have agreed to participate in research
* Affiliated to a social security scheme
* major

Exclusion Criteria:

* Diabetes , for diabetes induces accelerated formation of advanced glycation end products , which could then be a confounding factor in our study.
* Protected by law .
* minors
* pregnant women
* Matt or pigmented skin because the skin hyperpigmentation interfere with reading the skin fluorescence giving falsely elevated values .
* Having an aneurysm of the abdominal aorta known
* Suffering from a progressive neoplastic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Frammingham Score | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Belmokhtar K, Ortillon J, Jaisson S, Massy ZA, Boulagnon Rombi C, Doue M, Maurice P, Fritz G, Gillery P, Schmidt AM, Rieu P, Toure F. Receptor for advanced glycation end products: a key molecule in the genesis of chronic kidney disease vascular calcification and a potential modulator of sodium phosphate co-transporter PIT-1 expression. Nephrol Dial Transplant. 2019 Dec 1;34(12):2018-2030. doi: 10.1093/ndt/gfz012. PMID 30778553